CLINICAL TRIAL: NCT03310203
Title: The Relation Between Adiposity, Inflammation, Glycaemia and Iron Absorption: A Comparison Between Central and Peripheral Adiposity
Brief Title: The Relation Between Adiposity, Inflammation, Glycaemia and Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: ETH Zurich (Switzerland) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NUT:OO:23
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Iron Absorption
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Obese women: central obesity (Experimental): OGTT with iron
  Interventions: Diagnostic Test: Iron
- Obese women: peripheral obesity (Experimental): OGTT with iron
  Interventions: Diagnostic Test: Iron
- Lean women (Experimental): OGTT with iron
  Interventions: Diagnostic Test: Iron

INTERVENTIONS:
Diagnostic Test: Iron — Labelled iron
  Other Names: OGTT

SUMMARY:
A total of 126 premenopausal women (42 lean, 42 obese with central obesity, 42 obese with peripheral obesity) will be recruited. Anthropometric measurements and body composition using DEXA will be collected. Overnight fasted subjects will be asked to give baseline blood samples before consuming a meal containing 6 mg 57Fe in the form of FeSO4. Subjects will return after 14 days and a blood sample will be collected for measurement of isotopic enrichment into red blood cells, serving as well as a baseline for the OGTT. Subjects will then be asked to ingest a solution of glucose (50g) containing 100 mg of iron in the form of sodium ferrous citrate (SFC), after which blood samples will be collected 2 hours post iron and glucose load. All three blood samples collected at baseline, 2 weeks post labeled iron load, and 2 hours post glucose/iron load will be analyzed for their levels of iron, glycaemia and inflammatory parameters.

DETAILED DESCRIPTION:
1. Obese subjects with central and peripheral obesity

   During the first phase, overweight/obese subjects with a BMI 28-35 Kg/m2 will be invited to a screening. At the screening, anthropometrics (weight, height, waist circumference) and body composition (using BIA and DEXA) will be measured. Based on the subject's distribution of body fat, those who have a predefined % body fat between 45-55% will be invited to join the study and they would fall into one of the following two groups:
   * 42 subjects with >43% fat in the android sector (area from the pelvis to 20% of the distance between the pelvis and the neck cuts) according to the DEXA results (central adiposity) would be recruited
   * 42 subjects with <43% fat in the android sector according to DEXA (peripheral adiposity) would be recruited.
2. Lean subjects At the same time, anthropometric (weight, height, waist circumference) and body composition (using BIA and DEXA) measurement will be conducted on interested lean subjects (BMI 20-25).

Overnight fasted subjects:

At T0:

There will be a determination of the type and degree of obesity through the measurement of weight, height, BMI, and WC, followed by both BIA screening and DEXA scan to obtain a more detailed image about the status of the participant.

At T1:

A fasting blood sample of 10 ml (4 ml EDTA coated tubes, 6 ml uncoated tubes) will be drawn to measure the inflammatory status, glycaemia, and iron levels of the participant by determining CRP, alpha-glycoprotein, hepcidin, ferritin, TfR, TIBC, HbA1c, insulin, FPG, serum iron, CBC and lipid profile.

After this blood test, the subject will be given a meal including 57Fe (6 mg iron as FeSO4).

At T2:

A second venous blood sample of 10 ml (4 ml EDTA coated tubes, 6 ml uncoated tubes) will be drawn for analysis of hemoglobin and erythrocyte isotopic composition as well as for the determination of serum ferritin, transferrin receptor, C-reactive protein, alpha-glycoprotein and hepcidin.

At T3:

A third venous blood sample of 10 ml (4 ml EDTA coated tubes, 6 ml uncoated tubes) will be drawn to measure the level of glucose, insulin, TG, FFA, TIBC and serum iron. This blood test will be an indicator of the level of glycaemia and iron appearance in the blood of the subject through the earlier ingestion of OGTT and oral iron load.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* pregnant women lactating women

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Iron absorption | two weeks
  Labelled iron enrichment in red blood cells
Glycemic response | 2 hours
  oral glucose load

SECONDARY OUTCOMES:
Iron absorption | 2 hours
  serum iron concentration

CONTACTS AND LOCATIONS:
Overall Officials: Omar Obeid, PhD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided